CLINICAL TRIAL: NCT07286448
Title: Personalized Digital Training for COGnitive FITness in Mild Cognitive Impairment: the COG-FIT Pragmatic Trial
Brief Title: Personalized Digital Training for COGnitive FITness in Mild Cognitive Impairment
Acronym: COG-FIT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Giovanna Zamboni (Other)
Collaborators: IRCCS Fondazione Don Carlo Gnocchi - ONLUS, Milan (Unknown)
Responsible Party: Sponsor-Investigator, Giovanna Zamboni, Full Professor of Neurology at the Department of Biomedical, Metabolic and Neural Sciences of the University of Modena and Reggio Emilia, University of Modena and Reggio Emilia
Organization: University of Modena and Reggio Emilia (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14610/2025
Record Dates: First submitted 2025-12-02; First posted 2025-12-16 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-12

CONDITIONS: Mild Cognitive Impairment (MCI); Subjective Cognitive Decline (SCD)
Keywords: Mild Cognitive Impairment; Digital Therapeutics; Cognitive Rehabilitation; Patient Activation; Home-Based Intervention
MeSH Terms: conditions — Cognitive Dysfunction; Patient Participation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RICORDO - Digital Cognitive Rehabilitation (Experimental): Participants assigned to this arm will receive a 5-week personalized cognitive training program using the CE-marked digital therapeutic RICORDO. The intervention consists of 15 tablet-based home sessions (3 per week, 45 minutes each), tailored to the participant's cognitive profile and performance, and remotely monitored by clinicians via a web platform.
  Interventions: Device: RICORDO
- S.A.M.B.A. - Lifestyle Education Program (Active Comparator): Participants assigned to this arm will follow a 5-week home-based educational program called S.A.M.B.A., which includes 15 sessions (3 per week) using printed and video materials focused on socialization, healthy nutrition, physical activity, psychological well-being, and environmental stimulation. This arm is matched for contact time and format but does not include cognitive training.
  Interventions: Behavioral: S.A.M.B.A.

INTERVENTIONS:
Device: RICORDO — RICORDO is a CE-marked digital therapeutic for cognitive rehabilitation, delivered via tablet. The program consists of home-based sessions, each lasting approximately 45 minutes. Tasks are automatically adapted based on the participant's baseline cognitive profile and real-time performance. Clinicians remotely monitor adherence and adjust the prescription through a web platform.
  Arms: RICORDO - Digital Cognitive Rehabilitation
Behavioral: S.A.M.B.A. — S.A.M.B.A. (Socialisation, Alimentazione, Movimento, Benessere psicologico, Ambiente) is a structured, home-based lifestyle education program. Participants receive printed and video materials and complete sessions covering key domains of brain-healthy behavior. This arm is matched in duration and frequency to the experimental arm but includes no cognitive training.
  Arms: S.A.M.B.A. - Lifestyle Education Program

SUMMARY:
The goal of this clinical trial is to determine whether a home-based digital cognitive-training program called RICORDO can enhance patients' ability to manage their own health and daily life when they have Mild Cognitive Impairment (MCI) or Subjective Cognitive Decline (SCD) and are 50 years of age or older.

The main questions it aims to answer are:

Does using RICORDO for five weeks raise the Patient Activation Measure (PAM) score more than an at-home paper-and-video education program called S.A.M.B.A.?

Does RICORDO also improve cognition, everyday functioning, quality of life and mood compared with S.A.M.B.A.?

Researchers will compare individuals who train with RICORDO to those who follow S.A.M.B.A. to determine which approach is more effective.

Participants will be randomly assigned to one of the two groups and complete three 45-minute sessions per week at home for five weeks. They will also visit the clinic at the beginning and end of the program to complete questionnaires and take brief thinking tests.

DETAILED DESCRIPTION:
The COG-FIT study is a pragmatic, single-blind, randomized controlled trial designed to assess the effectiveness of RICORDO, a CE-marked digital cognitive rehabilitation intervention, in improving patient activation and autonomy in individuals with Mild Cognitive Impairment (MCI) and Subjective Cognitive Decline (SCD).

The study is sponsored by the University of Modena and Reggio Emilia and funded under the Italian National Recovery and Resilience Plan (PNC0000007 - FIT4MEDROB). It is a post-marketing clinical investigation of a certified medical device software, conducted in accordance with EU Regulation 2017/745.

Participants (n=100) will be recruited from two outpatient centres in Modena and Milan, Italy. Eligible individuals will be randomly assigned (1:1) to either:

RICORDO group: 15 home-based sessions (3/week, 45 minutes each) using a personalized digital training program delivered via tablet, guided by adaptive algorithms based on the patient's MoCA profile, baseline clinical information and performance over time.

Active control group (S.A.M.B.A.): 15 sessions with video and printed materials on lifestyle domains (Social interaction, Nutrition, Physical activity, Psychological well-being, Environment), matched for duration and frequency.

Primary and secondary outcome measures will be collected at baseline (T0) and after 5 weeks (T1) by blinded assessors. The primary endpoint is the change in Patient Activation Measure (PAM). Secondary endpoints include cognitive function (MoCA, CRIq), functional status (WHODAS 2.0), quality of life (EQ-5D-5L), and neuropsychiatric symptoms (STAI-Y, BDI-II, MBI-C). Usability (SUS) and technology acceptance (TAM) will be assessed in the RICORDO group at T1.

Participants' adherence will be tracked digitally (RICORDO) or via logbooks (S.A.M.B.A.), with weekly phone support. Data will be pseudonymized and entered into REDCap servers hosted in Italy, which are managed in accordance with GDPR and national privacy laws.

The study is powered to detect a mean PAM difference of 8.8 points (SD = 12) based on previous trials. With α = 0.05, power = 90%, and a 20% dropout rate, the total sample size is set at 100. Statistical analyses will be conducted on an intention-to-treat basis, with imputation of missing data and sensitivity checks.

No invasive procedures or pharmacological interventions are planned. All participants will provide informed consent. Risk is minimal due to the non-invasive nature of the intervention, and adverse events will be closely monitored.

The total duration of the study is 12 months, with 9 months of recruitment and a 5-week intervention per participant. Results will be disseminated through open-access publications, public events, and the project's website.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Mild Cognitive Impairment (MCI) based on Petersen (1999) and Winblad (2004), or Subjective Cognitive Decline (SCD) according to Jessen (2014)
* Mini-Mental State Examination (MMSE) > 18 and Clinical Dementia Rating (CDR) ≤ 1
* Age ≥ 50 years
* Formal education > 3 years
* Signed informed consent
* Stable neurotropic pharmacological therapy in the past 3 months (if applicable)
* Preserved mental capacity (i.e., not under legal guardianship or protective supervision)
* Preserved ability to understand and produce written and spoken Italian

Exclusion Criteria:

* Severe sensory or communication impairments
* Recent participation (< 3 months) in cognitive or rehabilitation programs
* Failure to provide or withdrawal of informed consent
* History or evidence of central nervous system disorders that may affect cognition and are unrelated to the study (e.g., major stroke, brain tumors, normal pressure hydrocephalus, traumatic brain injury)
* History or evidence of major psychiatric disorders
* Presence of medical conditions that may interfere with cognitive function (e.g., renal or hepatic failure, obstructive sleep apnea, hypothyroidism, vitamin B12 deficiency)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-11-28 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Patient Activation Measure | Baseline (T0) and 5 weeks (T1)
  The Patient Activation Measure (PAM) is a validated and highly reliable scale designed to assess a person's level of activation, defined as their ability to manage their own health and actively participate in care. The PAM identifies four progressive levels of activation: (1) awareness of the importance of one's role in managing health, (2) acquisition of the knowledge and confidence to take action, (3) initiation of health-related behaviors, and (4) consistent maintenance of those behaviors even under stress (Hibbard et al., 2004).

SECONDARY OUTCOMES:
Montreal Cognitive Assessment | Baseline (T0) and 5 weeks (T1)
  The MoCA is a brief cognitive screening tool used to detect mild cognitive impairment. It assesses multiple domains, including attention and concentration, executive functions, memory, language, visuoconstructional skills, abstract reasoning, calculation, and orientation. The test takes approximately 10 minutes to administer and has a maximum score of 30 points; scores of 26 or above are generally considered within the normal range. Tasks include the Trail Making Test, complex figure copying, object naming, word and sentence repetition, attention and verbal fluency tests, abstraction, and orientation questions. Each item is scored according to standardized criteria, allowing for reliable evaluation of a participant's cognitive performance.
Cognitive Reserve Index questionnaire | Baseline (T0) only
  The CRIq is a psychometric tool designed to assess the cumulative cognitive reserve developed across the lifespan. It evaluates three main domains: education, working activity, and leisure time, and provides an overall composite score of an individual's cognitive reserve. The CRIq is widely used in clinical and neuropsychological research to investigate the protective role of cognitive reserve in age-related cognitive decline and neurodegenerative diseases. Due to its simplicity, reliability, and validity, it is considered a useful tool in both clinical and epidemiological settings.
World Health Organization Disability Assessment Schedule 2.0 | Baseline (T0) and 5 weeks (T1)
  The WHODAS 2.0 is a standardized, cross-culturally applicable instrument developed by the World Health Organization to assess health and disability in the general adult population and in clinical settings. WHODAS 2.0 assesses functioning across six key domains: cognition, mobility, self-care, social interaction, daily activities, and participation in society. Grounded in the framework of the International Classification of Functioning, Disability and Health (ICF), it measures health and disability as a continuum, regardless of the underlying medical condition. WHODAS 2.0 is available in two main versions-a 36-item full form and a 12-item short form-administered via interview, self-report, or proxy. It provides a composite score reflecting the functional impact of different health conditions and supports monitoring and planning of healthcare interventions.
EuroQol-5 Dimension | Baseline (T0) and 5 weeks (T1)
  The EQ-5D-5L is a standardized and quick-to-administer instrument designed to assess health-related quality of life (HRQL) from the patient's perspective. It evaluates five key dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is rated across five severity levels, generating up to 3,125 unique health states and providing a detailed picture of an individual's health status. The EQ-5D-5L also includes a visual analogue scale (VAS) ranging from 0 (the worst imaginable health state) to 100 (the best imaginable health state), allowing patients to provide a global rating of their perceived health. Due to its simplicity and versatility, it is widely used in clinical practice, economic evaluations, and epidemiological research, enabling comparisons across conditions and populations.
State-Trait Anxiety Inventory Form Y | Baseline (T0) and 5 weeks (T1)
  The STAI-Y is a widely used psychometric instrument for assessing anxiety in adults and older adults. It includes two 20-item subscales that distinguish between state anxiety (S-Anxiety), a temporary emotional condition in response to situational stress, and trait anxiety (T-Anxiety), a stable tendency to perceive situations as threatening. The STAI-Y has been validated in older Italian populations, demonstrating high internal consistency and strong psychometric properties. Normative data are available for this population, supporting its use in clinical and research settings to identify anxiety levels that may negatively affect overall health, cognitive functioning, and quality of life in older adults.
Beck Depression Inventory | Baseline (T0) and 5 weeks (T1)
  The BDI is a 21-item self-report questionnaire designed to assess the presence and severity of depressive symptoms and attitudes. Originally developed by Beck in 1961, it takes approximately 10 minutes to complete and requires a basic reading level. The BDI demonstrates high internal consistency and robust psychometric properties across both psychiatric and general populations. It is one of the most widely used tools in clinical and research settings to screen for depression and monitor symptom severity over time.
Mild Behavioral Impairment Checklist | Baseline (T0) and 5 weeks (T1)
  The MBI-C is a specialized instrument designed to assess emergent neuropsychiatric symptoms in individuals aged 50 years and older, which may precede cognitive decline or dementia. It includes 34 items grouped into five domains: decreased motivation, emotional dysregulation, impulse control difficulties, socially inappropriate behaviour, and abnormal thoughts or perceptions. The MBI-C captures behavioural changes that persist for at least 6 months and represent a meaningful deviation from the individual's previous baseline. It can be completed by the patient, a knowledgeable informant, or a clinician. The tool is valuable for the early detection of dementia-related syndromes and for monitoring symptom progression over time.
System Usability Scale | 5 weeks (T1 only)
  The SUS is a widely used psychometric tool for evaluating users' perceived ease of use of a product, interface, or service. It consists of 10 items rated on a 5-point Likert scale (ranging from "strongly disagree" to "strongly agree") and yields a single composite score that reflects the overall perceived usability of the system.
Technology Acceptance Model | 5 weeks only (T1)
  TAM is a widely used psychometric framework for explaining and predicting user acceptance and usage of new technologies. It focuses on two key constructs: perceived usefulness and perceived ease of use, both of which influence users' attitudes toward the technology and their intention to use it. TAM has been validated in multiple settings and has demonstrated strong reliability and utility in forecasting the adoption of new technologies in workplace, healthcare, and educational contexts.

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliero Universitaria di Modena, Modena, Reggio Nell'Emilia (RE), Italy

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the study involves cognitively vulnerable individuals and data sharing could raise concerns about privacy and identifiability, even after pseudonymization. Additionally, the current ethics approval does not include provisions for external data sharing.